CLINICAL TRIAL: NCT01008046
Title: N-acetyl Cysteine Plus Clomiphene Citrate Versus Metformin and Clomiphene Citrate in Treatment of Clomiphene-resistant Polycystic Ovary Syndrome
Brief Title: N-acetyl Cysteine and Clomiphene Citrate or Metformin and Clomiphene Citrate for Women With CC Resistant Polycystic Ovary Syndrome (PCOS).
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Dr. Hatem Abu Hashim, Associate Prof. of OB/GYN, Mansoura Faculty of Medicine, Mansoura University.
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MU- 183; FMH-112-M
Record Dates: First submitted 2009-11-04; First posted 2009-11-05 (Estimated); Last update posted 2009-11-05 (Estimated); Status verified 2009-11

CONDITIONS: Polycystic Ovary Syndrome
Keywords: Polycystic ovary syndrome; clomiphene resistance; metformin; N-acetyl cysteine
MeSH Terms: conditions — Polycystic Ovary Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- combined N-acetyl cysteine - CC (Experimental): N-acetyl cysteine(1.8 g orally daily)for 5-6 weeks from the 1st day of spontaneous or induced menstruation followed by 100 mg CC for 5 days from day 3 of spontaneous or induced menstruation. With persistent anovulation,CC increased by 50 mg for the next cycle. Treatment continued for three successive cycles
  Interventions: Drug: combined N-acetyl cysteine -CC
- combined metformin-CC (Active Comparator): Patients received metformin HCl (1500 mg daily) for 5-6 weeks from the 1st day of spontaneous or induced menstruation, followed by 100 mg CC for 5 days starting from day 3 of spontaneous or induced menstruation. With persistent anovulation,CC increased by 50 mg for the next cycle. Treatment continued for three successive cycles.
  Interventions: Drug: combined metformin-CC

INTERVENTIONS:
Drug: combined N-acetyl cysteine -CC — N-acetyl cysteine(1.8 g orally daily)for 5-6 weeks from the 1st day of spontaneous or induced menstruation followed by 100 mg CC for 5 days from day 3 of spontaneous or induced menstruation. With persistent anovulation,CC increased by 50 mg for the next cycle. Treatment continued for three successive cycles
  Arms: combined N-acetyl cysteine - CC
Drug: combined metformin-CC — Patients received metformin HCl (1500 mg daily) for 5-6 weeks from the 1st day of spontaneous or induced menstruation, followed by 100 mg CC for 5 days starting from day 3 of spontaneous or induced menstruation. With persistent anovulation,CC increased by 50 mg for the next cycle. Treatment continued for three successive cycles
  Arms: combined metformin-CC

SUMMARY:
The purpose of this study is to compare and determine the efficacy of combined N-acetyl cysteine and clomiphene citrate(CC)with combined metformin and CC in infertile women with Polycystic ovary syndrome(PCOS)not responding to treatment with Clomiphene alone.

DETAILED DESCRIPTION:
In combined NAC-CC group group,patients received NAC (200 mg per sachet, SEDICO, Egypt) for 5-6 weeks from the 1st day of of spontaneous or induced menstruation (in a dose of 1.8 g orally in three divided doses, 3 sachets per dose). All patients in other group received metformin HCl (Cidophage®; Chemical Industries Development, Egypt), 500 mg thrice daily for 5-6 weeks from the 1st day of spontaneous or induced menstruation. Then after the end of this period, patients in either group received 100 mg CC (Clomid®; Global Napi Pharmaceuticals,Cairo, Egypt) for 5 days starting from day 3 of spontaneous or induced menstruation. With persistent anovulation, it was increased by 50 mg for the next cycle. Patients continued treatment for three successive cycles using the same protocol. NAC and metformin were stopped only when pregnancy was documented.

ELIGIBILITY:
Inclusion Criteria:

* CC resistant PCOS

Exclusion Criteria:

* Congenital adrenal hyperplasia
* Cushing syndrome
* Androgen secreting tumors

Ages: 20 Years to 36 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 192 (Actual)
Dates: Start 2007-04; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
Ovulation rate

SECONDARY OUTCOMES:
pregnancy rate

CONTACTS AND LOCATIONS:
Overall Officials: Hatem Abu Hashim, MD. MRCOG, Principal Investigator — Mansoura University Hospital; Kamal Anwar, MD, Study Chair — Mansoura University Hospital; Rafat Abd El-Fatah, MD, Study Director — Mansoura University Hospital
Locations (1):
- Mansoura University Hospitals,OB/GYN department, Al Mansurah, Dakahlia Governorate, Egypt

REFERENCES:
- [Background] Elnashar A, Fahmy M, Mansour A, Ibrahim K. N-acetyl cysteine vs. metformin in treatment of clomiphene citrate-resistant polycystic ovary syndrome: a prospective randomized controlled study. Fertil Steril. 2007 Aug;88(2):406-9. doi: 10.1016/j.fertnstert.2006.11.173. Epub 2007 Mar 1. PMID 17335818
- [Background] Rizk AY, Bedaiwy MA, Al-Inany HG. N-acetyl-cysteine is a novel adjuvant to clomiphene citrate in clomiphene citrate-resistant patients with polycystic ovary syndrome. Fertil Steril. 2005 Feb;83(2):367-70. doi: 10.1016/j.fertnstert.2004.07.960. PMID 15705376
- [Background] Siebert TI, Kruger TF, Steyn DW, Nosarka S. Is the addition of metformin efficacious in the treatment of clomiphene citrate-resistant patients with polycystic ovary syndrome? A structured literature review. Fertil Steril. 2006 Nov;86(5):1432-7. doi: 10.1016/j.fertnstert.2006.06.014. Epub 2006 Sep 27. PMID 17007847